CLINICAL TRIAL: NCT02000687
Title: Long Term Surveillance of Islet Transplant Recipients Following Complete Graft Loss
Status: Recruiting | Type: Observational
Sponsor: Rodolfo Alejandro (Other)
Responsible Party: Sponsor-Investigator, Rodolfo Alejandro, Professor of Medicine, University of Miami
Organization: University of Miami (Other)
Other Study IDs: 20080127
Record Dates: First submitted 2013-11-26; First posted 2013-12-04 (Estimated); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a single-center, prospective, open label study in islet transplant recipients following islet graft loss.

DETAILED DESCRIPTION:
After complete islet graft loss is determined, patient's maintenance immunosuppression (i.e. sirolimus, tacrolimus, MMF and/or Myfortic®) will be discontinued and they will be monitored for 10 years thereafter, for the appearance of allosensitization using panel reactive antibody (PRA) levels and monitor the persistence of elevated PRA levels. Primary objective is to determine the rate of allosensitization in patients 3 years after failed islet transplantation (i.e. stimulated c-peptide <0.3mg/mL) and monitor the persistence of elevated PRA levels (≥ 20%) at year 3, 6, and 9. Timing, frequency and level of change in PRA will be monitored after all immunosuppression is discontinued.

ELIGIBILITY:
Inclusion Criteria:

1. History of at least one islet alone transplant (ie islet transplant in the absence of any other organ transplant).

Exclusion Criteria:

1. Inability to provide written informed consent.
2. Mentally unstable and/or unable to comply with the procedures of the study protocol.
3. History of any solid organ transplant.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ages 18-75 years old that received at least one IT. Participants will be obtained from the pool of islet transplant recipients transplanted at the Diabetes Research Institute at the University of Miami, Miller School of Medicine.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2008-12; Primary Completion 2027-12 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
determine the rate of allosensitization in patients after failed islet transplantation | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Rodolfo Alejandro, MD, Principal Investigator — University of Miami
Locations (1):
- Diabetes Research Institute, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Rios P, Baidal D, Lemos J, Camhi SS, Infante M, Padilla N, Alvarez Gil AM, Fuenmayor V, Ambut J, Qasmi FA, Mantero AM, Cayetano SM, Ruiz P, Ricordi C, Alejandro R. Long-term Persistence of Allosensitization After Islet Allograft Failure. Transplantation. 2021 Nov 1;105(11):2490-2498. doi: 10.1097/TP.0000000000003635. PMID 33481552
- See also: Diabetes Research Institute clinical trials — https://diabetesresearch.org/dri-clinical-trials/